CLINICAL TRIAL: NCT05338970
Title: A Phase 3, Randomized, Open-label Study of Patritumab Deruxtecan Versus Platinum-based Chemotherapy in Metastatic or Locally Advanced Epidermal Growth Factor Receptor-mutated (EGFRm) Non-small Cell Lung Cancer (NSCLC) After Failure of Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) Therapy (HERTHENA-Lung02)
Brief Title: HERTHENA-Lung02: A Study of Patritumab Deruxtecan Versus Platinum-based Chemotherapy in Metastatic or Locally Advanced EGFRm NSCLC After Failure of EGFR TKI Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U31402-A-U301; 2021-005879-40 (EudraCT Number); jRCT 2021220002 (Other: JAPIC)
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Nonsquamous Non-small Cell Lung Cancer; EGFR L858R; EGFR Exon 19 Deletion
Keywords: Nonsquamous Non-small Cell Lung Cancer; EGFR L858R; EGFR exon 19 deletion; Patritumab deruxtecan; HER3-DXd; U3-1402
MeSH Terms: interventions — patritumab deruxtecan; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patritumab deruxtecan (Experimental): Participants who will be randomized to receive patritumab deruxtecan (HER3-DXd) 5.6 mg/kg q3W.
  Interventions: Drug: Patritumab Deruxtecan
- Platinum-based chemotherapy (Active Comparator): Participants who will be randomized to receive platinum-based chemotherapy for 4 cycles: pemetrexed plus either cisplatin or carboplatin. Participants without disease progression after 4 cycles of platinum plus pemetrexed therapy may continue treatment with maintenance pemetrexed with no restriction on the number of cycles.
  Interventions: Drug: Platinum-based chemotherapy

INTERVENTIONS:
Drug: Patritumab Deruxtecan — Intravenous administration, 5.6 mg/kg every 3 weeks (q3W)
  Other Names: HER3-DXd; U3-1402
  Arms: Patritumab deruxtecan
Drug: Platinum-based chemotherapy — Intravenous, pemetrexed 500 mg/m^2 plus either cisplatin (75 mg/m^2) or carboplatin (target area under the plasma concentration time curve of 5 [AUC5] by using the Calvert formula) q3W
  Arms: Platinum-based chemotherapy

SUMMARY:
Disease progression is typical for patients with epidermal growth factor receptor mutated (EGFRm) non-small cell lung cancer (NSCLC). Standard platinum-based chemotherapy offers limited efficacy and an unfavorable safety profile.There is an urgent need for more effective and tolerable therapies for patients with EGFRm NSCLC who have exhausted available targeted therapies. Clinical evidence suggest that patritumab deruxtecan constitutes a promising investigational therapy for patients with EGFRm NSCLC.

DETAILED DESCRIPTION:
Patritumab deruxtecan (HER3-DXd, U3-1402) is an antibody-drug conjugate (ADC) comprising an anti-HER3 mAb linked to a topoisomerase I inhibitor that is in clinical development for patients with NSCLC, metastatic breast cancer, and colorectal cancer.

The primary objective of the current study is to compare the efficacy of patritumab deruxtecan versus platinum-based chemotherapy, as measured by progression-free survival (PFS) and the key secondary endpoint of overall survival (OS), in participants with metastatic or locally advanced NSCLC with an EGFR-activating mutation (exon 19 deletion or L858R) after failure of third-generation (eg, osimertinib, lazertinib, aumolertinib, alflutinib) EGFR TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female subject aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
2. Has histologically or cytologically documented metastatic or locally advanced non-squamous NSCLC not amenable to curative surgery or radiation.
3. Has documentation of an EGFR-activating mutation detected from tumor tissue or blood sample: exon 19 deletion or L858R at diagnosis or thereafter.
4. Received 1 or 2 prior line(s) of an approved EGFR TKI treatment in the metastatic or locally advanced setting, which must include a third -generation EGFR TKI
5. May have received either neoadjuvant and/or adjuvant treatment if progression to metastatic or locally advanced disease occurred at least 12 months after the last dose of such therapy and subsequently experienced disease progression on or after third-generation EGFR TKI treatment administered in the metastatic or locally advanced setting.
6. Has not received any other prior systemic therapies in the metastatic or locally advanced setting (including chemotherapy, immunotherapy etc) (even if administered in combination with EGFR TKI).
7. Has documentation of radiographic disease progression while receiving or after receiving a third generation EGFR TKI for metastatic or locally advanced disease.
8. Has at least 1 measurable lesion as per RECIST v1.1 by Investigator assessment.
9. Is willing to have a tumor biopsy or provide recently obtained tumor tissue.
10. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at Screening.
11. Has adequate bone marrow reserve and organ function based on local laboratory evaluation within 14 days prior to randomization:

    * Platelet count: ≥100,000/mm^3 or ≥100 × 10^9/L within 14 days prior to the assessment of platelet count during the Screening Period
    * Absolute neutrophil count: ≥1500/mm^3 or ≥1.5 × 10^9/L within 14 days prior to the assessment of absolute neutrophil count during the Screening Period
    * Hemoglobin (Hgb): ≥9.0 g/dL within 14 days prior to the assessment of hemoglobin during the Screening Period
    * Creatine clearance (CrCl): CrCl ≥45 mL/min calculated by using the Cockcroft-Gault equation or measured CrCl
    * Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT): AST/ALT ≤3× Upper limit of normal (ULN)
    * Total bilirubin (TBL): TBL ≤1.5 × ULN
    * Serum albumin: ≥2.5 g/dL
    * Prothrombin time (PT) or Prothrombin time-International normalized ratio (PT-INR) and activated partial thromboplastin time (aPTT)/partial thromboplastin time (PTT): ≤1.5 × ULN, except for participants receiving coumarin-derivative anticoagulants or other similar anticoagulant therapy who must have PT-INR within therapeutic range as deemed appropriate by the Investigator

Exclusion Criteria:

1. Has any previous histologic or cytologic evidence of small cell OR combined small cell/non-small cell disease in the archival tumor tissue or pretreatment tumor biopsy, or squamous NSCLC histology
2. Has any history of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis), has current ILD, or is suspected to have such disease by imaging during Screening
3. Has clinically severe respiratory compromise (based on the Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to the following:

   * Any underlying pulmonary disorder, restrictive lung disease, or pleural effusion
   * Any autoimmune, connective tissue, or inflammatory disorders where there is documented, or a suspicion of pulmonary involvement at the time of Screening
   * OR prior complete pneumonectomy
4. Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to randomization
5. Has any history of or evidence of current leptomeningeal disease
6. Has evidence of clinically active spinal cord compression or brain metastases, defined as being symptomatic and untreated, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
7. Any prior treatment with any agent including an antibody drug conjugate (ADC) containing a chemotherapeutic agent targeting topoisomerase I, human epidermal growth factor receptor 3 (HER3) antibody, and any systemic therapies (other than EGFR TKIs) in the metastatic/locally advanced setting, including chemotherapy or any other systemic therapy in combination with an EGFR TKI
8. Has history of other active malignancy within 3 years prior to randomization, except for adequately resected nonmelanoma skin cancer, adequately treated intraepithelial carcinoma of the cervix, and any other curatively treated in situ disease
9. Has uncontrolled or significant cardiovascular disease prior to randomization
10. Has active hepatitis B and/or hepatitis C infection, such as those with serologic evidence of active viral infection within 28 days of randomization
11. Has a known human immunodeficiency virus (HIV) infection that is not well controlled
12. Has clinically significant corneal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) Based on RECIST v1.1 | Baseline up to approximately 49 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to the earlier of the dates of the first documentation of objective progression of disease or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline up to approximately 49 months
  Overall survival (OS) is defined as the time from the date of randomization to the date of death due to any cause.
Progression-free Survival (PFS) as Assessed by Investigator Review Based on RECIST v1.1 | Baseline up to approximately 49 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to the earlier of the dates of the first documentation of objective progression of disease or death due to any cause.
Progression-free Survival (PFS) as Assessed by Local Standard Clinical Practice | Baseline up to approximately 49 months
  Progression-free survival (PFS) by local standard clinical practice is defined as the time from date of randomization to the documented progression on the first new anticancer therapy (if administered) or death due to any cause, whichever occurred first.
Objective Response Rate (ORR) as Assessed by BICR and Investigator Review Based on RECIST v1.1 | Baseline up to approximately 49 months
  Objective response rate (ORR) is defined as the proportion of participants who have a confirmed best overall response (BOR) of complete response (CR) or partial response (PR).
Duration of Response (DoR) as Assessed by BICR and Investigator Review Based on RECIST v1.1 | Baseline up to approximately 49 months
  Duration of response (DoR) is defined as the time from the first documentation of objective response (CR or PR) to the earlier of the dates of the first documentation of objective progression of disease or death due to any cause.
Clinical Benefit Rate (CBR) as Assessed by BICR and Investigator Review Based on RECIST v1.1 | Baseline up to approximately 49 months
  Clinical benefit rate (CBR) will be assessed by BICR and Investigator based on RECIST v1.1. CBR is defined as the proportion of participants who have a confirmed BOR of CR, PR, or stable disease (SD) that lasts for at least 180 days.
Disease Control Rate (DCR) as Assessed by BICR and Investigator Review Based on RECIST v1.1 | Baseline up to approximately 49 months
  Disease control rate (DCR) is defined as the proportion of participants who have a confirmed BOR of CR, PR, or SD.
Time to Response (TTR) as Assessed by BICR and Investigator Review Based on RECIST v1.1 | Baseline up to approximately 49 months
  Time to response (TTR) is defined as the time from the date of randomization to the date of the first documentation of response (CR or PR) that is subsequently confirmed.
Intracranial PFS as Assessed by BICR | Baseline up to approximately 49 months
  Intracranial PFS is defined as the time from the date of randomization to the earlier of the dates of the first documented radiographic intracranial disease progression or death, whichever comes first, as assessed by BICR per CNS-RECIST, in participants with CNS lesion(s) at baseline by BICR per CNS-RECIST.
Mean Change from Baseline in Non-small Cell Lung Cancer - Symptom Assessment Questionnaire | Baseline up to approximately 49 months
  The NSCLC-SAQ will assess disease-related symptom change in patients with NSCLC.
Mean Change from Baseline in Patient's Global Impression of Change | Baseline up to approximately 49 months
  The PGI-C is a 7-point scale depicting a participant's rating of overall improvement.
Mean Change from Baseline in Patient's Global Impression of Severity | Baseline up to approximately 49 months
  The PGI-S is a one-item questionnaire that contains six response options.
Mean Change from Baseline in Patient's Global Impression of Treatment Tolerability | Baseline up to approximately 49 months
  The PGI-TT will capture the patient's overall impression of treatment tolerability.
Mean Change from Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline up to approximately 49 months
  The EORTC-QLQ-C30 will assess the patient's overall quality of life (QoL).
Mean Change from Baseline in EuroQol Questionnaire-5 dimensions-5 levels (EQ-5D-5L) | Baseline up to approximately 49 months
  The EQ-5D-5L is a standardized instrument that will be used for measuring generic health status required for health technology assessments.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline up to approximately 49 months
  TEAEs will be graded by using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
Percentage of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) | Baseline up to approximately 49 months
  The immunogenicity of patritumab deruxtecan will be confirmed by assessing the anti-drug antibodies.
Percentage of Participants Who Have Treatment-emergent ADA | Baseline up to approximately 49 months
  The immunogenicity of patritumab deruxtecan will be confirmed by assessing the anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo; Clinical Scientist, Study Chair — Daiichi Sankyo
Locations (179):
- United States (23):
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Highlands Oncology, Springdale, Arkansas
  - City of Hope, Duarte, California
  - Moores Cancer Center at the UC San Diego Health, La Jolla, California
  - Scripps MD Anderson Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente - Vallejo Medical Center, Vallejo, California
  - Innovative Clinical Research Institute, Whittier, California
  - Sarah Cannon/Florida Cancer Specialists - FCS South, Port Charlotte, Florida
  - Emory University, Atlanta, Georgia
  - St Luke's Cancer Institute, Boise, Idaho
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack Meridian Health-Southern Ocean Medical Center, Manahawkin, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Australia (6):
  - The Chris O'Brien Lifehouse, Camperdown
  - St George Public Hospital, Kogarah
  - Liverpool Hospital, Liverpool
  - Austin Hospital, Melbourne
  - St John of God Subiaco Hospital, Subiaco
  - Princess Alexandra Hospital, Woolloongabba
- Austria (5):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Klinikum Klagenfurt Pulmologie, Klagenfurt
  - Karl Landsteiner Institut fur Lungenforschung und pneumologische Onkologie c/o Klinik Floridsdorf, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
  - AZ Sint Maarten Mechelen, Mechelen
  - AZ Delta, Roeselare
- William Osler Health System - Brampton Civic Hospital, Brampton, Canada
- China (26):
  - Peking University Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - University of Electronic Science Technology of China UESTC - Sichuan Cancer Hospital Institute Sichuan Provincial Tumor Hospital, Chengdu
  - National Cancer Center Hospital East, Chibi
  - Fujian Medical University - Union Hospital Foochow Christian Union Hospital, Fuzhou
  - Guangdong Academy of Medical Science (GAMS) - Guangdong Provincial Peoples Hospital, Guangzhou
  - The First Affiliated Hospital Sun-Yat-Sen University, Guangzhou
  - Pecking University Third Hospital, Haidian
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou
  - Zhejiang Cancer hospital, Hangzhou
  - Harbin Medical University - Tumor Hospital The Third Affiliated Hospital, Harbin
  - The First Affiliated Hospital - Anhui Medical University Dept of Medical Oncology, Hefei
  - Henan Provincial Peoples Hospital, Henan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - Lin Yi Cancer Hospital, Linyi
  - General Hospital of Eastern Theater Command, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Fudan University - Shanghai Cancer Center FUSCC, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - The First Hospital of China Medical University, Shenyang
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Huazhong University of Science and Technology - Tongji Medical College - Tongji Hospital TJH, Wuhan
  - The First Affiliate Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- France (10):
  - Hopital Morvan CHU de Brest, Brest
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Montpellier Cancer Institute ICM, Montpellier
  - Institut Curie, Paris
  - APHP - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire (CHU) de Rennes - Hopital de Pontchaillou, Rennes
  - Institut de Cancrologie de lOuest ICO, Saint-Herblain
  - Gustave Roussy, Villejuif
- Germany (10):
  - Universitaetsklinikum Essen, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - IKF Krankenhaus Nordwest, Frankfurt am Main
  - Asklepios Fachklinik Muenchen-Gauting, Gauting
  - Universitatsklinik Giessen und Marburg, Giessen
  - LungenClinic Grosshansdorf, Großhansdorf
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - LKI Lungenfachklinik Immenhausen, Immenhausen
  - Klinikverbund Allgaeu, Kempten
  - Pius-Hospital Oldenburg, Oldenburg
- Hong Kong (4):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - University of Hong Kong/Queen Mary Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
- Italy (11):
  - IRCCS Istituto Oncologico Giovanni Paolo II, Bari
  - University G. D'Annunzio Chieti, Chieti
  - Ospedale San Luca, Lucca
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Santa Maria della Misericordia, Perugia
  - IFO Regina Elena, Roma
  - IRCCS Humanitas Research Hospital, Rozzano
  - ASST Sette Laghi, Varese
- Japan (22):
  - Hyogo Cancer Center, Akashi
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Kansai Medical University Hospital, Hirakata
  - Iwakuni Clinical Center, Iwakuni
  - Izumi City General Hospital, Izumi
  - Kanazawa University Hospital, Kanazawa
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - Kurume University Hospital, Kurume
  - Matsusaka Municipal Hospital, Matsusaka
  - NHO Shikoku Cancer Center, Matsuyama
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Ōsaka-sayama
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Sendai Kousei Hospital, Sendai
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (6):
  - Netherlands Cancer Institute, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - St. Jansdal Ziekenhuis, Harderwijk
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Norway (3):
  - Akershus University Hospital, Nordbyhagen
  - Oslo University Hospital-The Norwegian Radium Hospital, Oslo
  - Stavanger University Hospital, Stavanger
- Poland (3):
  - II Klinika Chorob Pluc i Gruzlicy, Bialystok
  - Onko-Centrum Sp. z o.o., Lublin
  - Med Polonia Sp. z o.o., Poznan
- Portugal (4):
  - Centro Clinico Champalimaud, Lisbon
  - Instituto Portugues de Oncologio de Lisboa, Lisbon
  - Centro Hospitalar Universitario do Porto - Hospital de Santo Antonio, Porto
  - Centro Hospitalar de Vila Nova de Gaia - Espinho, Porto
- Singapore (4):
  - National University Cancer Institute National University Hospital, Singapore
  - National Cancer Centre Singapore NCCS, Singapore
  - Tan Tock Seng Hospital, Singapore
  - ICON Cancer Centre, Singapore
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- Spain (12):
  - Hospital Teresa Herrera C.H.U.A.C., A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Complejo Hospitalario Materno-Insular - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Malaga, Málaga
  - Hospital Univeritario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
- Switzerland (2):
  - Kantonsspital Graubuenden - Hauptstandort, Chur
  - Kantonsspital Winterthur KSW, Winterthur
- Taiwan (6):
  - E-Da Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital NCKUH, Tainan
  - National Taiwan University Hospital NTUH, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou Branch, Taoyuan District
- United Kingdom (9):
  - University Hospital Birmingham NHS Trust, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Cancer Centre, Leeds
  - University Hospitals of Leicester, Leicester
  - Barts and The London NHS Trust - St Bartholomew s hospital - PET CT Centre, London
  - The Royal Marsden Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie Hospital, Manchester
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Mok T, Janne PA, Nishio M, Novello S, Reck M, Steuer C, Wu YL, Fougeray R, Fan PD, Meng J, Sternberg DW, Esker S, Yu HA. HERTHENA-Lung02: phase III study of patritumab deruxtecan in advanced EGFR-mutated NSCLC after a third-generation EGFR TKI. Future Oncol. 2024 May;20(15):969-980. doi: 10.2217/fon-2023-0602. Epub 2023 Dec 14. PMID 38095056
- [Derived] Yu HA, Goto Y, Hayashi H, Felip E, Chih-Hsin Yang J, Reck M, Yoh K, Lee SH, Paz-Ares L, Besse B, Bironzo P, Kim DW, Johnson ML, Wu YL, John T, Kao S, Kozuki T, Massarelli E, Patel J, Smit E, Reckamp KL, Dong Q, Shrestha P, Fan PD, Patel P, Sporchia A, Sternberg DW, Sellami D, Janne PA. HERTHENA-Lung01, a Phase II Trial of Patritumab Deruxtecan (HER3-DXd) in Epidermal Growth Factor Receptor-Mutated Non-Small-Cell Lung Cancer After Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and Platinum-Based Chemotherapy. J Clin Oncol. 2023 Dec 10;41(35):5363-5375. doi: 10.1200/JCO.23.01476. Epub 2023 Sep 10. PMID 37689979